CLINICAL TRIAL: NCT06171581
Title: Effect of Stress Ball Use on Anxiety Level During Endometrial Biopsy Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Yeliz DİNÇER, Dr, Principle İnvestigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 'ZonguldakBEU'
Record Dates: First submitted 2023-10-25; First posted 2023-12-14 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Biopsy Wound; Endometrial Hyperplasia; Endometrial Neoplasms
Keywords: stress ball; endometrial biopsy; women
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized control study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental-stress ball (Experimental): The study is planned to consist of two groups as experimental and control.
  No intervention will be given to the control group.
  Interventions: Other: stress ball
- no intervention- none (Experimental): The study is planned to consist of two groups as experimental and control.
  No intervention will be given to the control group.
  Interventions: Other: control

INTERVENTIONS:
Other: stress ball — In the study, the experimental group was given a round, compressible ball for stress ball application and it was planned to squeeze this ball in their hands as often as they wanted during anaesthesia and endometrial biopsy application. The endometrial biopsy procedure is a procedure that usually takes between 8-10 minutes. The results will be evaluated considering these average times. As it is foreseen that individuals may experience the most intense anxiety and stress during anaesthesia and biopsy, it was preferred to cover this time period.
  Other Names: experimental group- stress ball
  Arms: experimental-stress ball
Other: control — In the study, the no intervention group ( control group) will receive no intervention and blood pressure and stress measurements will be made with routine care and nursing interventions.
  Other Names: no intervention-control
  Arms: no intervention- none

SUMMARY:
The aim of this study is to determine the effect of stress ball application on the anxiety level during the endometrial biopsy procedure.

This research is planned as a randomised controlled study. Place and time of the research: The research is planned with patients who will undergo endometrial biopsy procedure in Zonguldak Obstetrics and Gynecology Hospital affiliated to the Ministry of Health.

While there are various experimental studies in the literature on the effect of stress ball on anxiety during many painful procedures, there is no study in the literature on the effect of stress ball on anxiety level during endometrial biopsy procedure (Akarsu, Kuş & Akarsu 2021, Genç 2021Nurdina, Anggraini & Novyanda 2022, Srivarsan, Sridevi & Preetha 2021, Yanks et al. 2018,) In this study, it was aimed to evaluate the effect of stress ball application on anxiety level during endometrial biopsy procedure

DETAILED DESCRIPTION:
Endometrial biopsy is a simple, inexpensive and effective method to rule out endometrial cancer.

Endometrial biopsy is the gold standard method in the diagnosis of endometrial pathologies and is widely used in gynaecological practice. Although endometrial biopsy is a common gynaecological procedure, its psychological effects have not been emphasised. In particular, the potential stress before and during the procedure, exposure to the test and the waiting time for the biopsy result have been mostly ignored. Patients with bleeding in the postmenopausal period already present to the physician with anxiety, and when it is stated that a biopsy should be taken for diagnosis, their anxiety increases due to both the procedure itself and the possibility of an unfavourable outcome at the end of the procedure.

While there are various experimental studies in the literature on the effect of stress ball on anxiety during many painful procedures, there is no study in the literature on the effect of stress ball on anxiety level during endometrial biopsy procedure .In this study, it was aimed to evaluate the effect of stress ball application on anxiety level during endometrial biopsy procedure.

ELIGIBILITY:
Inclusion Criteria:

EXPERIMENT GROUP

* Willingness to participate in the research
* 18 years of age or older
* Reading and writing Turkish
* No active mental illness preventing data collection
* No impediment to squeezing the ball
* No emergency and risky situation that will prevent data collection during the process CONTROL GROUP
* Willingness to participate in the research
* 18 years of age or older
* Reading and writing Turkish
* No active mental illness preventing data collection
* No emergency and risky situation that will prevent data collection during the process

Exclusion Criteria:

INTERVENTION GROUP

* Not willing to participate in the research
* Under 18 years of age
* Not knowing how to read and write Turkish
* Having an active mental illness that prevents data collection
* Having an obstacle to squeezing the ball
* The development of an urgent and risky situation that will prevent data collection during the process CONTROL GROUP
* Not willing to participate in the research
* Under 18 years of age
* Not knowing how to read and write Turkish
* Having an active mental illness that prevents data collection
* The development of an urgent and risky situation that will prevent data collection during the process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
"State and Trait Anxiety Scale" | before and after the biopsy procedure(1-2 minutes before and 1-2 minutes after biopsy procedure)
  The state and trait anxiety scale consists of two parts and contains a total of 40 questions. The first 20 questions of the scale measure state anxiety, and the last 20 questions measure trait anxiety. The results of the state anxiety section of the scale will be used in this research. The State Anxiety Scale requires the individual to describe how he or she feels at a particular moment and under certain circumstances.
"Visual Analogue Scale (VAS)" ( min 0- max 10) | before and after the biopsy (1-2 minutes before and 1-2 minutes after biopsy procedure)
  It constitutes another parameter for measuring the stress level.
blood pressure ( systolic and diastolic) mm/ hg | before and after the biopsy (1-2 minutes before and 1-2 minutes after biopsy procedure)
  The aim is to determine the changes caused by stress on blood pressure before and after the procedure.

IPD SHARING:
Plan to Share IPD: Yes
The study is planned to be completed within 1 year and published as a publication within 3 years.
Supporting Information: Study Protocol
Time Frame: It is planned to be published within 3 years
Access Criteria: The study is planned to be published openly.